CLINICAL TRIAL: NCT07137065
Title: A Multilevel Intervention for Low Back Pain Management in Primary Care: An Effectiveness-implementation Hybrid Study
Brief Title: A Multilevel Intervention for Low Back Pain Management in Primary Care
Acronym: PRIME Back
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guillaume Christe (Other)
Collaborators: Haute Ecole de Santé Vaud (HESAV), Lausanne, Switzerland (Unknown); University of Geneva, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Guillaume Christe, Associate Professor, Haute Ecole de Santé Vaud
Organization: Haute Ecole de Santé Vaud (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRIME_2025_08_08; PT0043_222873 (Other Grant/Funding Number: SNFS)
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain
Keywords: Primary care; Guidelines implementation
MeSH Terms: conditions — Low Back Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: This study uses an effectiveness-implementation hybrid design (type 1), which prioritizes the evaluation of clinical effectiveness while collecting detailed information on the implementation process. The study is a cluster randomized controlled trial, with the unit of randomization being quality circles of general practitioners (GPs) affiliated with a care network in the French-speaking part of Switzerland. A total of 20 quality circles will be randomized into intervention and control arms. Each quality circle includes multiple GP practices, and approximately 100 GPs will participate in total.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All outcome measures will be directly recorded in Redcap by the participants (no outcome assessor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRImary care MultilEvel intervention for low back pain (PRIME) (Experimental): For general practitioners in this arm, they will receive 2 x 1 hour of training, will have access to trained physiotherapists and will use a dedicated clinical pathway based on risk of chronicity.
  Interventions: Behavioral: PRImary care MultilEvel intervention for low back pain (PRIME)
- Usual Care (Active Comparator): General practitioners in this arm will continue to practice as usual.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: PRImary care MultilEvel intervention for low back pain (PRIME) — The multilevel intervention includes four main components:
  1. GP training. GPs will receive training to improve their confidence in LBP guidelines, diagnostic triage and best practice. Furthermore, they will be trained to provide both general and cognitive reassurance to patients, use a stratified care strategy and improve interprofessional communication. 2. Reminders. GPs will receive regular reminders by email to reinforce the integration of high-value care into practice. 3. Patient education. GPs will reassure patients, help them understand their LBP in the initial consultation and target unhelpful beliefs about LBP. 4. Clinical pathway. The clinical pathway includes a gradual stratified care pathway based on risk factors for chronicity. The core interventions of this 3-step clinical pathway are education and self-management, individual sessions with a trained physiotherapist, and multidisciplinary group management. GPs remain free to make all clinical decisions.
  Other Names: Healthcare professional training; Reminders; Patient education; Stratified care
  Arms: PRImary care MultilEvel intervention for low back pain (PRIME)
Other: Usual Care — In this arm, general practitioners will treat their patients as usual. They can prescribed any treatment or diagnostic tests to their patients.
  Arms: Usual Care

SUMMARY:
Low back pain is the leading cause of disability worldwide and one of the main reasons for consulting in primary care. This project aims to improve the management of people with low back pain in primary care through an innovative intervention developed in collaboration with general practitioners, physiotherapists, and occupational therapists.

The main objective is to test the effectiveness of a multilevel intervention designed to improve the care pathway for individuals with low back pain consulting their general practitioner. The intervention supports healthcare professionals in adopting practices based on current guidelines, promotes patient education, and offers an interprofessional care pathway tailored to each person's needs and profile.

The study will include over 100 general practitioners in French-speaking Switzerland, randomly assigned to either the intervention group or the control group (usual care). Around 500 patients will be followed according to their doctor's approach. Their progress will be monitored over 12 months using questionnaires and administrative data.

This project addresses an urgent need to improve the care pathway in primary care. It will rigorously assess the effectiveness of this new care approach and explore the barriers and facilitators to its integration into daily practice, taking into account the experiences of both healthcare professionals and the people concerned.

DETAILED DESCRIPTION:
Using an effectiveness-implementation hybrid type I design, this study aims to test the effectiveness of a multilevel intervention in primary care for patients with LBP and investigate the implementation processes.

The primary objectives are to test the effectiveness of a multilevel intervention in primary care for patients with low back pain (PRIME: PRImary care MultilEvel intervention for low back pain) compared with usual care in terms of: (1.1) Cost-effectiveness (system-level) (1.2) Imaging prescription rate (practitioner-level); (1.3) Self-reported back-related disability (patient-level).

Secondary objectives are:

2.1 To evaluate the effectiveness of the PRIME intervention on opioid prescription rate and sick leave days prescription by general practitioners (practitioner-level) 2.2 To evaluate the effectiveness of the PRIME intervention on pain intensity, work participation, health-related quality of life, global perceived change, Pain Self-Efficacy, Fear Avoidance Beliefs, and beliefs about LBP (patient-level) 2.3 To evaluate the effectiveness of the training on clinicians' beliefs about LBP and confidence in treating patients with LBP (practitioner-level)

As an effectiveness-implementation hybrid design type 1 study, implementation process outcomes are secondary objectives. These include: (3.1) evaluating the acceptability, appropriateness, feasibility, fidelity and adoption of the multilevel intervention among general practitioners, physiotherapists and occupational therapists; (3.2) exploring barriers and facilitators to the implementation of the multilevel intervention among healthcare practitioners; (3.3) exploring the experience of a biopsychosocial 2-day experiential workshop among trained physiotherapists; (3.4) exploring the experience and acceptability of the multilevel intervention among patients.

The study is a cluster randomized controlled trial, with the unit of randomization being quality circles of general practitioners affiliated with a care network in the French-speaking part of Switzerland. A total of 20 quality circles will be randomized into intervention and control arms. Each quality circle includes multiple general practitioner practices, and approximately 100 general practitioners will participate in total.

General practitioners in the intervention group will receive a multilevel intervention including: general practitioners training, reminders, tools for patients education and a dedicated clinical pathway. The clinical pathway includes a gradual stratified care pathway based on risk factors for chronicity. The core interventions of this 3-step clinical pathway are education and self-management, individual sessions with a trained physiotherapist, and multidisciplinary group management. Physiotherapists providing individual sessions in the intervention group will all have participated in a two-day workshop to improve their knowledge of good clinical practice and develop their competence to manage risk factors of chronicity within a biopsychosocial framework. They will be trained to address unhelpful beliefs and avoidance behaviors through good communication and gradual exposure exercises, as improving unhelpful beliefs and reducing kinesiophobia are important mediators of successful rehabilitation. If general practitioners recommend multidisciplinary group management, patients will receive a comprehensive assessment of risk factors and tailored education by an experienced occupational therapist. If this confirms the need for multidisciplinary group management, patients will receive a structured outpatient multidisciplinary group rehabilitation for LBP that specifically targets physical and psychological factors.

The clinical pathway provides advice to general practitioners at three stages:

In the first consultation, general practitioners will screen for red flags, reassure and explain LBP to patients with the above-mentioned resources, and prescribe medication if needed. They will also decide whether the patient needs to immediately start physiotherapy sessions with a trained physiotherapist.

Ten days after the first consultation, patients will receive an SMS/email directing them to an online questionnaire that assesses risk factors of chronicity (Start Back Tool) and their ability to work. General practitioners will automatically receive via email a summary of the risk of chronicity (low, medium or high) and the patient ability to work. The email will only communicate the current state of the patient and the general practitioner is free to decide whether to follow the clinical pathway recommendation, as independence of practice is also important for implementation. If the patient has already been prescribed trained physiotherapy, it is suggested that nothing is changed at that time (10 days), independent of the level of risk. Coordination of care with the physiotherapist is strongly advised in this case. In case physiotherapy has not yet been prescribed, general practitioners are advised the following:

(i) If the patient is able to work normally and has a low risk of chronicity, he or she should continue to self-manage and the general practitioner should decide to organize a follow-up meeting based on the patient needs; (ii) If the patient has a medium or high risk of chronicity, or is still not able to work normally because of LBP, the general practitioner is advised to prescribe 6 sessions of trained physiotherapy (with the possibility to prescribe additional sessions in the future).

At 6 weeks after the first consultation, patients will receive another SMS/email with the same questionnaire to fill out, and general practitioners will receive the automated email again. At 6 weeks, general practitioners will be advised the following:

(i) If the patient is able to work normally and has a low risk of chronicity, it is probable that the patient has recovered. Therefore, no new treatment should be started and physical activity should be promoted. A follow-up consultation can be organized if needed.

(ii) If the patient is able to work normally and has a medium risk of chronicity, prescription of trained physiotherapy would be advised for 6 sessions if not yet started. If physiotherapy was already started and the patient is improving, 6 additional sessions could be offered at this stage based on patient and physiotherapist reports; (iii) If the patient is not able to work normally or has high risk of chronicity, general practitioners would be advised to offer a comprehensive assessment of risk factors and tailored education by a specialized occupational therapist. If this confirms the need for multidisciplinary treatment, multidisciplinary management could be started.

Importantly, for patients that have already started physiotherapy, physiotherapists and general practitioners are advised to work together to coordinate care, as interprofessional collaboration was highlighted to be a critical point in the pilot study.

The primary effectiveness outcomes include patient-reported back-related disability (measured by the Roland-Morris Disability Questionnaire), the proportion of patients referred for spinal imaging within three months, and the incremental cost per quality-adjusted life year (QALY) gained. Secondary patient outcomes include pain intensity, health-related quality of life, work participation, pain self-efficacy, fear avoidance beliefs, general beliefs about LBP, and global perceived improvement. Practitioner-level outcomes include opioid and sick leave prescription rates, as well as changes in GP confidence and beliefs about LBP.

General practitioners in the control group will have no specific training or intervention and will treat patients according to their usual practice.

Implementation outcomes are evaluated using both quantitative and qualitative methods. These include the acceptability, appropriateness, feasibility, adoption, and fidelity of the intervention among general practitioners, physiotherapists, and occupational therapists. The experience of the physiotherapists who complete a two-day biopsychosocial training workshop is also explored. Patient perspectives on the acceptability of the intervention will be collected through interviews or focus groups.

Patients data collection will occur at baseline and at 10 days, 6 weeks, 3, 6, 9, and 12 months. Patients complete questionnaires online via REDCap at each time point. Administrative data and prescribing behavior are also collected to complement self-reported outcomes. General practitioners will complete questionnaires before and after training and at the end of the recruitment period. Focus groups and interviews with healthcare professionals and patients will be recorded, anonymized, transcribed, and analyzed using thematic analysis.

The target sample size is at least 500 patients, with approximately 25 per cluster. Recruitment may exceed this number to ensure that a minimum of 200 patients per group complete the 6-month follow-up. The study has been powered to detect a minimal clinically important difference of 2.5 points on the Roland-Morris scale, assuming a standard deviation of 6 and an intracluster correlation coefficient (ICC) of 0.05. Analyses will be conducted according to the intention-to-treat principle, using linear and generalized linear mixed models to account for clustering. Cost-effectiveness will be assessed from both the healthcare payer and societal perspectives using the EQ-5D-5L.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting their participating general practitioner for a primary concern of LBP (with or without leg pain)
* Above 18 years old

Exclusion Criteria:

* If they had consulted their general practitioner for a primary concern of LBP in the past 3 months, as care was already started prior to the study.
* Unable to give consent (eg. cognitive impairment)
* Unable to access comfortably an electronic device to answer the questionnaires (smartphone, computer)
* Unable to answer questionnaires in French
* Known pregnancy
* Have had back surgery in the last 6 months
* Any specific cause of LBP (e.g. inflammatory arthritis, malignancy, infection, fracture, cauda equina syndrome).
* a major strength deficit (M3 and below) due to radiculopathy or have to be referred directly to emergency or a specialist because of that. As specific causes of LBP may be unknown at the first consultation in primary care, patients with a confirmed diagnosis of specific LBP could be excluded post-allocation by an independent doctor that is part of the Data Monitoring Committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean incremental cost per quality-adjusted life-year (QALY) calculated using the EQ-5D-5L questionnaire | 0-12 months period after enrolment
  Primary system-level outcome measures will be the mean incremental cost per quality-adjusted life-year (QALY) calculated using the EQ-5D-5L questionnaire from a healthcare payer and a societal perspective
Back-related imaging rate (%) among patients with low back pain | 0-6 months period after enrolment
  The primary practitioner-level outcome measure will be the back-related imaging rate (%) among patients with LBP during 6 months after the primary consultation.
Self-reported back-related disability measured with the Roland Morris Disability Questionnaire | 6 months after enrolment
  The primary patient-level outcome will be self-reported back-related disability measured with the Roland Morris Disability Questionnaire (RMDQ) six months after the initial general practitioner consultation

SECONDARY OUTCOMES:
Pain intensity with the Numerical Rating Scale | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  Secondary patient-level outcome measures will be pain intensity with the Numerical Rating Scale (NRS)
Health-related quality of life (HRQL) with the EQ-5D-5L questionnaire | 3, 6, 12 months after enrolment
  Secondary patient-level outcome measures will be health-related quality of life (HRQL) with the EQ-5D-5L questionnaire
Work participation with the Work Productivity and Activity Impairment Questionnaire (WPAI) | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  Work participation will be measured with the Work Productivity and Activity Impairment Questionnaire (WPAI) (patient-level outcome)
Pain Self-Efficacy with the Pain Self Efficacy Questionnaire short form (PSEQ-2) | 6 weeks and 6 months after enrolment
  Pain Self-efficacy will be measured by the Pain Self Efficacy Questionnaire short form (PSEQ-2) (patient-level outcome)
Fear of movement | 6 weeks and 6 months after enrolment
  Fear of movement will be measured with the Brief Screening Questions on Fear of movement (Kent al. 2014) (patient level outcome)
Catastrophization | 6 weeks and 6 months after enrolment
  Catastrophization will be measured with the Brief Screening Questions on Fear of movement (Kent al. 2014) (patient level outcome)
Anxiety | 6 weeks and 6 months after enrolment
  Anxiety will be measured with the single question from the Orebro short form questionnaire (patient-level outcome)
Depression | 6 weeks and 6 months after enrolment
  Depression will be measured with the single question from the Orebro short form questionnaire (patient-level outcome)
Beliefs about back pain | 6 weeks and 6 months after enrolment
  Beliefs about back pain will be measured with the 10-item Back-PAQ questionnaire (patient-level outcome)
Short question about confidence to perform activities people value | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  Based on the advice of our patient partner, we added this question (patient-level outcome):
  How confident are you in your back's ability to support you in your daily activities?
Short question about capacity to perform activities people value | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  Based on the advice of our patient partner, we added this question (patient-level outcome):
  To what extent can you perform the daily activities you value?
Number of patients receiving an opioid prescription | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  To collect data on opioid prescription rate, we will ask if they had been prescribed opioid for their LBP. In addition, we will ask patients in the informed consent the possibility to request healthcare costs to their insurance, including prescription rate of opioid.
Dose of opioid prescription per patient | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  For opioids, we will also determine the differences between groups in Morphine Milligram Equivalent (MME) per patient (practitioner-level outcome).
Back-specific imaging rate over 12 months | 0-12 months periods after enrolment
  Back-related imaging rate (%) among patients with LBP during 12 months after the primary consultation.
Total number of imaging exams between groups | 0-6 months period
  We will compare the total number of imaging exams between groups
Medication prescription | 10 days, 6 weeks, 3 months, 6 months, 9 months, 12 months after enrolment
  We will collect the number of medication prescribed (practitioner-level outcome)
Confidence in treating patients with LBP | Baseline, directly after healthcare practitioner training (average of 3 months after baseline), 6 months after healthcare practitioner training (average of 9 months after baseline).
  Confidence in treating patients with LBP will be measured with four questions from Smucker et al. 1998 (practitioner-level outcome)
Beliefs about back pain | Baseline, directly after healthcare practitioner training (average of 3 months after baseline), 6 months after healthcare practitioner training (average of 9 months after baseline).
  Belief about back pain will be measured with the 10-item Back-PAQ questionnaire (practitioner-level outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Christe, PhD, Principal Investigator — Haute Ecole de Santé Vaud
Locations (2):
- Switzerland (2):
  - Geneva, Geneva, Canton of Geneva
  - Vaud, Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Yes
All data that can be shared (informed consent, ethical aspects) will be shared. These data will be made public at the end of project on the Swiss-based data management portal OLOS. The data set will be assigned a globally unique and persistent identifier (PID) to make it easily findable.
  The data set will be thoroughly described, including description of the metadata, the protocol and procedures to collect the data, the license of the data and how it can be (re)used. The documents describing the data set and data will always have the PID of the data set and will be fully accessible.
Supporting Information: Study Protocol
Time Frame: After the study completion